CLINICAL TRIAL: NCT04476979
Title: Comparison of Tocilizumab Plus Dexamethasone vs. Dexamethasone for Patients With Covid-19
Acronym: TOCIDEX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200375-TOCIDEX; 2020-001246-18 (EudraCT Number)
Record Dates: First submitted 2020-07-16; First posted 2020-07-20 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Coronavirus Infection; SARS (Severe Acute Respiratory Syndrome); Virus Diseases; Coronaviridae Infections; Nidovirales Infections; RNA Virus Infections; Respiratory Tract Infections; Respiratory Tract Disease
MeSH Terms: conditions — Coronavirus Infections; Severe Acute Respiratory Syndrome; Virus Diseases; Coronaviridae Infections; Nidovirales Infections; RNA Virus Infections; Respiratory Tract Infections; Respiratory Tract Diseases | interventions — tocilizumab; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone (Active Comparator): Dexamethasone : 10 mg once daily for the first five days (day 1 to day 5) then 5 mg per day for up to 5 days, 2.5mg per day for up to 4 days (or until oxygen supply independency if sooner)
  Interventions: Drug: Dexamethasone
- Dexamethasone + Tocilizumab (Experimental): Dexamethasone : 10 mg once daily for the first five days (day 1 to day 5) then 5 mg per day for up to 5 days, 2.5mg per day for up to 4 days (or until oxygen supply independency if sooner)
  +Tocilizumab 8mg/kg D1 and if no response (No decrease of oxygen requirement) a second fixed dose of 400mg wil be administered at D3
  Interventions: Drug: Tocilizumab; Drug: Dexamethasone

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab 8mg/kg D1 and if no response (No decrease of oxygen requirement) a second fixed dose of 400mg wil be administered at D3
  Arms: Dexamethasone + Tocilizumab
Drug: Dexamethasone — Dexamethasone : 10 mg once daily for the first five days (day 1 to day 5) then 5 mg per day for up to 5 days, 2.5mg per day for up to 4 days (or until oxygen supply independency if sooner)

SUMMARY:
The overall objective of the study is to determine the therapeutic effect and tolerance of Tocilizumab combined with Dexamethasone in patients with moderate, severe pneumonia or critical pneumonia associated with Coronavirus disease 2019 (COVID-19).

Tocilizumab (TCZ) is an anti-human IL-6 receptor monoclonal antibody that inhibits signal transduction by binding sIL-6R and mIL-6R.

The study has a cohort multiple Randomized Controlled Trials (cmRCT) design. Randomization will occur prior to offering Dexamethasone alone or Dexamethasone +Tocilizumab administration to patients enrolled in the CORIMUNO-19 cohort.

Tocilizumab will be administered to consenting adult patients hospitalized with COVID-19 either diagnosed with moderate or severe pneumonia requiring no mechanical ventilation or critical pneumonia requiring mechanical ventilation.

Patients who will chose not to receive Tocilizumab will receive standard of cares.

Outcomes of Tocilizumab-treated patients will be compared with outcomes of standard of care (including Dexamethasone) treated patients

ELIGIBILITY:
Inclusion Criteria:

1. Patients included in the CORIMUNO-19 cohort
2. Patients belonging to the following group:

   * Requiring ≥ 3L/min of oxygen
   * WHO progression scale = 5
   * No NIV or High flow

Exclusion Criteria:

* Patients with exclusion criteria to the CORIMUNO-19 cohort.
* Known hypersensitivity to Tocilizumab or DXM or to any of their excipients.
* Pregnancy
* Current documented bacterial infection not controlled by antibiotics.
* certain evolving viral diseases (especially active herpes, chickenpox, shingles),
* psychotic states still not controlled by treatment,
* live vaccines in the previous 4 weeks,
* Active tuberculosis or disseminated strongyloidiasis
* Patient with any of following laboratory results out of the ranges detailed below at screening should be discussed depending of the medication:

  * Absolute neutrophil count (ANC) ≤ 1.0 x 109/L
  * Haemoglobin level: no limitation
  * Platelets (PLT) < 50 G /L
  * SGOT or SGPT > 5N

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-11 (Actual)

PRIMARY OUTCOMES:
Survival without needs of invasive ventilation at day 14 | day 14
  Survival without needs of invasive ventilation at day 14. Thus, events considered are mechanical (invasive) ventilation or death. A new DNR order will be considered as an event at the actual date of care limitation.

SECONDARY OUTCOMES:
WHO progression scale at day 7 and 14 | day 7 and day 14
  WHO progression scale:
  Uninfected; non viral RNA detected: 0 Asymptomatic; viral RNA detected: 1 Symptomatic; Independent: 2 Symptomatic; Assistance needed: 3 Hospitalized; No oxygen therapy: 4 Hospitalized; oxygen by mask or nasal prongs: 5 Hospitalized; oxygen by NIV or High flow: 6 Intubation and Mechanical ventilation, pO2/FIO2>=150 OR SpO2/FIO2>=200: 7 Mechanical ventilation, (pO2/FIO2<150 OR SpO2/FIO2<200) OR vasopressors (norepinephrine >0.3 microg/kg/min): 8 Mechanical ventilation, pO2/FIO2<150 AND vasopressors (norepinephrine >0.3 microg/kg/min), OR Dialysis OR ECMO: 9 Dead: 10
Overall survival at 14, 28, 60 and 90 days | 14, 28, 60 and 90 days
  Overall survival
Cumulative incidence of discharge alive at 14 and 28 days | 14 and 28 days
  Cumulative incidence of discharge alive
Survival without needs of mechanical ventilation at day 1 | day 1
  Survival without needs of mechanical ventilation at day 1. New DNR order (if given after the inclusion of the patient) will be considered as an event at the date of the DNR.
Cumulative incidence of oxygen supply independency at 14 and 28 days | 14 and 28 days
  Cumulative incidence of oxygen supply independency
Survival without needs of ventilator utilization at day 14 | 14 days
  Survival without needs of ventilator utilization (including non-invasive ventilation and Optiflow) at day 14

CONTACTS AND LOCATIONS:
Locations (1):
- CH Andrée Rosemon, Cayenne, French Guiana

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Hermine O, Mariette X, Porcher R, Djossou F, Nguyen Y, Arlet JB, Savale L, Diehl JL, Georgin-Lavialle S, Cadranel J, Pialoux G, Lacombe K, Mekinian A, Gros H, Lescure X, Ghosn J, Coupez E, Grapin K, Rapp C, Michel M, Lecapitaine AL, Michot JM, Costedoat-Chalumeau N, Nguyen LBL, Semerano L, Raffi F, Aguillar C, Rouzaud C, Gottenberg JE, Hansmann Y, Bienvenu B, London J, Fantchou FS, Ackermann F, Gros A, Morel A, Gambier N, Sene D, Megarbane B, Azoulay E, Bureau S, Dougados M, Emmerich J, Fartoukh M, Guidet B, Humbert M, Mahevas M, Pene F, Schlemmer F, Pourcher-Martinez V, Tibi A, Baron G, Perrodeau E, Baron S, Steg G, Yazdapanah Y, Simon T, Resche-Rigon M, Tharaux PL, Ravaud P. Tocilizumab plus dexamethasone versus dexamethasone in patients with moderate-to-severe COVID-19 pneumonia: A randomised clinical trial from the CORIMUNO-19 study group. EClinicalMedicine. 2022 Mar 25;46:101362. doi: 10.1016/j.eclinm.2022.101362. eCollection 2022 Apr. PMID 35350097